CLINICAL TRIAL: NCT03427931
Title: Continuous Glucose Monitoring in Islet Transplant Recipients
Brief Title: CGM Use in Islet Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20294
Record Dates: First submitted 2017-12-29; First posted 2018-02-09 (Actual); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Islet Transplantation; Type1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Islet Transplantation; Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Glucose Monitor (CGM) (Experimental): Study subjects will collect Continuous Glucose Monitor data by wearing the device at home a minimum of 28 days but may continue for up to 3 months.
  Interventions: Other: Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Other: Continuous Glucose Monitor (CGM) — Study subjects will collect Continuous Glucose Monitor data for a minimum of 28 days but may continue for up to 3 months.

SUMMARY:
A study assessing glucose variability in subjects with Type 1 Diabetes who have had islet transplant.

DETAILED DESCRIPTION:
Subjects who have an Islet Transplantation may have several outcomes including time when insulin is not required followed in some cases by additional insulin for glucose control as patients get further away from transplantation. It is unclear what role automated insulin delivery systems will have in addressing glucose variability in this group of patients who may have some amount of islet function. As a precursor to understanding ways in which automated insulin delivery systems may need to be adapted, we propose to gather data on glucose variability and insulin regimens in individuals who have undergone an islet transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus
* Recipient of Islet Transplantation
* Age 18 or older
* Females, not currently know to be pregnant
* Demonstration of proper mental status and cognition for the study
* Understanding and willingness to follow the protocol and informed consent form
* Access to the internet and willingness to upload data during the study, including use of personal laptop

Exclusion Criteria:

* Pregnancy and intent to become pregnant during trial
* Use of acetaminophen (such as Tylenol)
* Current enrollment in another intervention clinical trial that affects glucose variability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A Brown, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitor (CGM)
Started | 7
Completed | 5
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Glucose Monitor (CGM)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] — Population: Available data at baseline.
  percentage of glycosylated hemoglobin
    number analyzed (Participants) | 5
    (all) | 6.9 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Time in Range 70-180 mg/dL by CGM
Description: Descriptive analysis for CGM use measuring percentage time in range of glucose between 70-180 mg/dL
Time Frame: 28-90 days
Population: Participants with available CGM data for analysis.
Measure: Mean (Standard Deviation); unit: percentage of CGM readings 70-180mg/dL
Arm/Group | Continuous Glucose Monitor (CGM)
Number analyzed (Participants) | 5
percentage of CGM readings 70-180mg/dL | 77 (12)

2. Secondary Outcome: Percentage Time in Range <70 mg/dL by CGM
Description: Descriptive glycemic analyses based on CGM data with glucose range <70 mg/dL
Time Frame: 28-90 days
Measure: Mean (Standard Deviation); unit: percentage of CGM readings <70mg/dL
Arm/Group | Continuous Glucose Monitor (CGM)
Number analyzed (Participants) | 5
percentage of CGM readings <70mg/dL | 3.6 (3.2)

ADVERSE EVENTS:
Time Frame: During use of study equipment up to 3 months
Arm/Group | Continuous Glucose Monitor (CGM)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03427931/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03427931/ICF_001.pdf